CLINICAL TRIAL: NCT04671940
Title: RECUT PLUS: Exploratory Study of Clonal Evolution in Cancer for Patients Undergoing Transoral Robotic Surgery for Radiation Exposed Residual/reCurrent Tumours of the Upper Aerodigestive Tract
Brief Title: Exploratory Study of Clonal Evolution in Cancer for Patients Undergoing Transoral Robotic Surgery for Radiation Exposed Residual/reCurrent Tumours of the Upper Aerodigestive Tract
Acronym: RECUT Plus
Status: Recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Biomedical Research Centre (Unknown); Oracle Cancer Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: CCR 5263
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort: Patients who have previously had radiotherapy and then have had their local residual/recurrent disease managed with salvage TORS at the Royal Marsden Hospital will be eligible for inclusion. They will be informed of the RECUT+ study by a member of their usual care team at RMH during their routine outpatient appointments for follow up of their H&N cancer.
  Potential participants will be asked to consent to provide blood/saliva sample for germline DNA and for permission for their original tumour biopsy sample and their residual/recurrent resection to undergo DNA analysis. Where patients have returned to their referring institution and are no longer under active regular follow up at RMH, a research pack will be sent to the patient via post and email. This pack will contain the Cover Letter, the Participant Information Sheet and the Informed Consent Form. It will also contain a saliva collection tube, buccal swab, blood tubes and instructions for how to provide blood/saliva samples.
  Interventions: Other: DNA Analysis
- Prospective Cohort: Patients who have previously had radiotherapy and then are due to have their local residual/recurrent disease managed with salvage transoral robotic surgery at the Royal Marsden Hospital (RMH) will be approached prior to their salvage surgery at a routine outpatient appointment. They will be asked to consent to provide blood/saliva sample for germline DNA pre and post operatively. They will also be asked for permission for their original tumour biopsy sample and their residual/recurrent resection to undergo DNA analysis
  Interventions: Other: DNA Analysis

INTERVENTIONS:
Other: DNA Analysis — Molecular analysis includes DNA analysis on the blood/saliva and on the cancer specimens from the biopsies & subsequent resections

SUMMARY:
Radical radiotherapy for head and neck squamous cell cancer (HNSCC) can be administered to primary disease with curative intent. Residual disease, recurrence or further tumours may subsequently occur in this irradiated field. It is unknown whether these cancers reflect primary resistance or represent the evolution of resistance on treatment.

Understanding this could allow stratification of patients to more effective primary treatments, such as transoral robotic surgery, or help tailor systemic therapies for these cancers in previously irradiated fields.

RECUT+ is an exploratory molecular analysis study to assess the selective impact of radiation therapy on HNSCC.

Participants will be recruited from the Royal Marsden Hospital (RMH), Chelsea, a tertiary referral H&N cancer unit in London, UK, specialising in transoral robotic surgery.

Retrospective participants will be identified from previous Head and neck MDT lists at RMH.

Prospective participants will be screened for by the RECUT+ team during the weekly H&N MDT meetings at the Royal Marsden Hospital (RMH).

Blood/saliva samples will be collected pre operatively (prospective participants) and post operatively (retrospective and prospective participants) for germline and circulating tumour DNA analysis.

Biopsy samples from the original cancer and resected specimens from the post radiotherapy residual/recurrent/new primary disease will undergo molecular analysis to assess for any selective impact of radiotherapy on these further tumours.

ELIGIBILITY:
Inclusion criteria

* Aged over 18
* Previous H&N cancer treated with radiotherapy.
* Undergoing TORS as part of their management for residual, recurrent or new primary H&N cancer.

Exclusion criteria

* Where TORS is used in a diagnostic setting only
* Nasopharyngeal and thyroid head and neck cancers
* Where no tissue specimens are available from the recurrent/residual/secondary tumour for the retrospective cohort

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing transoral robotic surgery for radiation exposed residual/recurrent/new primary tumours of the upper aerodigestive tract.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2026-10-07 (Estimated); Study Completion 2026-10-07 (Estimated)

PRIMARY OUTCOMES:
Identification of resistant sub clones in post radiotherapy tumour samples | Within 1 year of surgery & receipt of blood/saliva and tissue samples
  Identification of resistant sub clones in post radiotherapy tumour samples

SECONDARY OUTCOMES:
Identification of differences in sub clonal architecture of H&N SCC before and after radiotherapy. | Within 1 year of surgery & receipt of blood/saliva and tissue samples
  Identification of differences in sub clonal architecture of H&N SCC before and after radiotherapy.
Identification of differences in mutational signatures between the primary disease and resistant sub clones. | Within 1 year of surgery & receipt of blood/saliva and tissue samples
  Identification of differences in mutational signatures between the primary disease and resistant sub clones.
Identification of loss of heterozygosity at the HLA loci in resistant sub clones | Within 1 year of surgery & receipt of blood/saliva and tissue samples
  Identification of loss of heterozygosity at the HLA loci in resistant sub clones
Disease-specific and overall survival at 5 years related to identified molecular characteristics. | 5 years following the date of surgery of the final participant recruited.
  Disease-specific and overall survival at 5 years related to identified molecular characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Vinidh Paleri, Principal Investigator — The Royal Marsden Hospital NHS Foundation Trust
Locations (1):
- The Royal Marsden Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT04671940/Prot_000.pdf
  • Informed Consent Form (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/40/NCT04671940/ICF_001.pdf